CLINICAL TRIAL: NCT00671008
Title: Efficacy of Glycaemic Control of Biphasic Insulin Aspart (NovoMix® 30) or Insulin Detemir (Levemir®) in Patients With Type 1 or 2 Diabetes Mellitus
Brief Title: Observational Study of Patients Using NovoMix® 30 or Levemir® for Treatment of Type 1 or Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1964
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: biphasic insulin aspart 30
- B
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoMix® 30
  Groups: A
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Groups: B

SUMMARY:
This trial is conducted in Europe.

The aim of this observational study is to evaluate the glycaemic control in patients with type 1 or 2 diabetes using NovoMix® 30 or Levemir® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 diabetes, including newly diagnosed
* Age: Levemir® above 6 years
* Age: Novomix® above 18 years

Exclusion Criteria:

* Current treatment with NovoMix® 30 or Levemir®

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 and Type 2 Diabetes Mellitus
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Glycaemic control as measured by HbA1c | After 24 weeks

SECONDARY OUTCOMES:
Percentage of subjects to reach HbA1c below 7.0% and =6.5% | After 24 weeks
Percentage of subjects on once vs twice daily injections of Levemir® or NovoMix® 30 | After 24 weeks
The effect on glycamic control as measured by FPG | After 24 weeks
The effect on glycamic control as measured by PG profile | After 24 weeks
Change in body weight | After 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Sarajevo, Bosnia and Herzegovina

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com